CLINICAL TRIAL: NCT00909740
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of MEGF0444A, Administered Intravenously to Patients With Advanced Solid Tumors
Brief Title: A Study of the Safety and Pharmacokinetics of MEGF0444A Administered to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEF4693g
Record Dates: First submitted 2009-05-20; First posted 2009-05-28 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Solid Cancers
Keywords: Solid Tumor; Cancer
MeSH Terms: conditions — Neoplasms | interventions — parsatuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MEGF0444A

INTERVENTIONS:
Drug: MEGF0444A — Intravenous escalating dose

SUMMARY:
This is a Phase I, first-in-human, open-label, dose-escalation study of MEGF0444A administered by IV infusion to patients with advanced solid tumors for whom standard therapy either does not exist or has proven to be ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable, or metastatic solid malignancy that has progressed on, or failed to respond to regimens or therapies known to provide clinical benefit

Exclusion Criteria:

* Inadequate hematologic and organ function
* Anti-cancer therapy within 4 weeks prior to initiation of study treatment
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia
* Active infection or autoimmune disease
* Pregnancy (positive pregnancy test) or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05-22 (Actual); Primary Completion 2011-10-26 (Actual); Study Completion 2011-10-26 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Days 1-21 of cycle 1
Incidence, nature, relatedness, and severity of adverse events | Day 1 to study completion

SECONDARY OUTCOMES:
Pharmacokinetic parameters including total exposure, minimum and maximum serum concentration, clearance, and volume of distribution | Following administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Louie Naumovski, M.D., Ph.D., Study Director — Genentech, Inc.